CLINICAL TRIAL: NCT05206110
Title: Low Dose Versus Normal Dose Ketorolac for Postoperative Pain After Prostatectomy and Hysterectomy: a Double-blind Randomized Controlled Non-inferiority Trial
Brief Title: Low Dose Versus Normal Dose Ketorolac for Postoperative Pain After Prostatectomy and Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principle Investigator, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: f/2021/129
Record Dates: First submitted 2022-01-07; First posted 2022-01-25 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Surgery
Keywords: Ketolorac; Dosage
MeSH Terms: interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients participating in the study, the surgeons, the researchers assessing the different outcome parameters and the data managers will all be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peri- and postoperative 10 mg Ketolorac (Experimental): Patients undergoing LAVH, RARP or TLH will receive dosages of 10 mg ketolorac (IV).
  Interventions: Drug: 10 mg IV ketorolac
- Peri- and postoperative standard-dose 30 mg Ketolorac (Active Comparator): Patients undergoing LAVH, RARP or TLH will receive standard dosages of 30 mg ketolorac (IV).
  Interventions: Drug: 30 mg IV ketorolac

INTERVENTIONS:
Drug: 10 mg IV ketorolac — Patients undergoing LAVH, RARP or TLH will receive half an hour before the end of surgery, 10 mg ketorolac (IV). Also, 10 mg IV ketorolac will be given 8h and 16h after the surgery
  Arms: Peri- and postoperative 10 mg Ketolorac
Drug: 30 mg IV ketorolac — Patients undergoing LAVH, RARP or TLH will receive half an hour before the end of surgery, 30 mg ketorolac (IV). Also, 30 mg ketorolac will be given 8h and 16h after the surgery
  Arms: Peri- and postoperative standard-dose 30 mg Ketolorac

SUMMARY:
A monocenter, prospective, double-blind, randomized controlled non-inferiority trial will be designed to investigate if ketorolac 10 mg is as effective for pain relief as the standard dose of 30 mg in patients undergoing robot assisted radical prostatectomy (RARP) or hysterectomy by laparoscopic assisted vaginal hysterectomy (LAVH) or total laparoscopic hysterectomy (TLH). It is hypothesised that the postoperative pain score at rest at 8 hours after surgery when receiving ketolorac 10 mg is non-inferior to the pain score at rest when receiving ketolorac 30mg.

DETAILED DESCRIPTION:
Ketorolac, a non-steroidal anti-inflammatory drug (NSAID), is a commonly used and effective drug for moderate to severe postoperative pain. It is widely prescribed as one of the first steps in acute and postoperative pain since decades. Because of its non-opioid character, this type of drug is safe concerning the risk of addiction and respiratory depression in the postoperative setting, but other side-effects are well known.

Gastro-intestinal (GI) haemorrhage is the most feared complication. The risk of a GI-bleeding increases with age, higher doses and longer duration of therapy. Decrease in renal function seems less important than always assumed. Feldman et al proved that developing renal failure with the use of NSAIDs was rather rare (1,1%) and similar for ketorolac as for opioids. Nonetheless, the risk again increased in a linear fashion with the duration of use. Especially for the postoperative and trauma patient, the fear of platelet inhibition and subsequent bleeding has dominated restriction of its use. Other adverse effects of ketorolac, i.e. cardiovascular toxicity, asthma, allergic reaction, etc., are usually less of a concern for the physician.

In an attempt to reduce these unwanted side effects but still have the benefit of its highly effective analgesic activity, patients should be given the lowest effective dose. Several studies have already demonstrated that ketorolac analgesic efficacy at 10 mg is similar to that at higher doses due to a ceiling effect. Unfortunately, none of the published trials investigated pain scores of the alternative dose beyond 6 hours. Based on the pharmacokinetics of ketorolac, it is possible that the lower dose will loose its analgesic effect after a shorter period. To investigate whether this alternative dose of ketorolac will preserve its analgesic efficacy up to eight hours postoperative, the primary goal of this study will be the pain score after 8 hours, right before the next dose of ketorolac.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years
* Patients undergoing RARP, LAVH or TLH
* ASA 1-3
* Scheduled as inpatient surgery (at least 1 night)
* Body weight > 60 kg

Exclusion Criteria:

* Refusal of the patient
* Cognitive impairment or no understanding of the Dutch language
* Allergy for salicylates or NSAID
* Pregnancy
* Active or history of peptic ulcer disease
* History of gastro-intestinal hemorrhage or perforation
* History of gastric bypass
* History of renal disease with creatinine > 1 mg/dl
* Haematological disease
* Tromboctopenia < 150000 / µl
* Current anticoagulant use
* Current clopidogrel use
* History of substance abuse or use of medication with a suppressive effect on the central nervous system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain at rest 8 hours after surgery: Numeric Rating Scale (NRS) | At 8 hours after surgery
  Pain at rest 8 hours after surgery (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)

SECONDARY OUTCOMES:
Pain at rest at PACU, 2, 4, 6, 12, 16 and 24 hours after surgery: Numeric Rating Scale (NRS) | At PACU, 2, 4, 6, 12, 16 and 24 hours after surgery
  Pain at rest at PACU, 2, 4, 6, 12, 16 and 24 hours after surgery (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Pain at movement at PACU, 2, 4, 6, 8, 12, 16 and 24 hours after surgery: Numeric Rating Scale | At PACU, 2, 4, 6, 8, 12, 16 and 24 hours after surgery
  Pain at movement at PACU, 2, 4, 6, 12, 16 and 24 hours after surgery (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Piritramide consumption at PACU (mg) | At PACU until 2 hours after surgery
  Mean total postoperative intravenous piritramide consumption at PACU (milligram)
Piritramide consumption first 24 hours postoperative (mg): PCIA pump | First 24 hours after surgery
  Total amount of intravenous piritramide used in the first 24h postoperative. Use of piritramide will be objectified by a patient controlled intravenous analgesia (PCIA) pump. Information on piritramide consumption will be extracted from the PCIA-system and analyzed using 4-hour intervals.
Quality of sleep during the first postoperative night: Numeric Rating Scale | First postoperative night
  Quality of sleep during the first postoperative night, as measured by an 11-point NRS (where 0 = no sleep at all, and 10 = sleeping very well)
Patient satisfaction: Numeric Rating Scale | 1week postoperatively assessed with telephone-call
  Overall patient satisfaction with pain therapy, as assessed with an 11-point NRS scale (where 0 = not satisfied at all and 10 = extremely satisfied).
Global Surgical Recovery Index | Before surgery (baseline) and 1 week postoperatively assessed with telephone-call
  General health status at that moment, as assessed with a scale (where 0=worst imaginable health status, and 100 = best imaginable health status)
EQ-5D | Before surgery (baseline) and 1 week postoperatively assessed with telephone-call
  Quality of life concerning mobility, self-care, pain/discomfort and anxiety/depression, as assessed with a score (where 0 = lowest quality of life, and 1 = highest quality of life)
Adverse effects of ketorolac use or suspected by the use of ketorolac | During study completion, i.e. 1 week after the surgery
  Possible adverse effects related to ketolorac are: GI-bleeding, acute kidney failure (defined as an increase in serum creatinine by 1,5), postoperative bleeding (defined as the necessity of packed cells transfusion or surgical relook), allergic reaction and asthma exacerbation.
Fear of the surgical procedure: Surgical fear questionnaire | Before surgery (baseline)
  Fear of the surgical procedure using an 8-item Surgical Fear Questionnaire.
Expected pain after surgery: Numeric Rating Scale | Before surgery (baseline)
  Expected pain after surgery measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Pain before surgery: Numeric Rating Scale | Before surgery (baseline)
  Pain before surgery measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No